CLINICAL TRIAL: NCT04920760
Title: The Effect of Vitamin A Supplementation on Disease Improvement of Children With Moderate to Severe COVID-19.
Brief Title: Vitamin A Supplementation in Children With Moderate to Severe COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyede Sedigheh Hamzavi, Assistant Professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 99-01-14-23475
Record Dates: First submitted 2021-06-09; First posted 2021-06-10 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: vitamin A; inflammation; pediatrics
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Intervention Model Description: The current phase II, prospective, single-center, single-blinded, randomized placebo-controlled trial, will compare the standard care alone (as the control arm) or in combination with ˝vitamin A supplementation˝ (as the intervention arm) with an allocation ratio of 1:1 in a parallel-group design.
Who Masked: Participant
Masking Description: Participants, laboratory technicians, and statisticians will be blinded to the study arm allocation. Investigators and the ICU medical staff, however, will be unblinded due to the nature of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants receiving standard treatment alone.
- Vitamin A (Experimental): Participants receiving standard treatment with an additional vitamin A supplementation.
  Interventions: Dietary Supplement: Vitamin A supplement

INTERVENTIONS:
Dietary Supplement: Vitamin A supplement — The supplementation protocol will be the additional care established by World Health Organization (WHO) and the United Nations International Children ʹs Fund (UNICEF) for measles (1998)(i.e. of 200,000 IU, or 50,000-100,000 IU for children > 1 or for infants of < 1 year of age, respectively).
  Arms: Vitamin A

SUMMARY:
Severe acute respiratory syndrome (SARS)-like coronavirus 2 (Sars-CoV-2) pandemia is considered to be the current major global health issue. With no specific treatment or vaccine known to be licensed, empowering the immune system to overcome the inflammatory status associated with the late stages of the disease, particularly by anti-inflammatory nutrients, is of great concern.

Effective in reducing both the morbidity and mortality of respiratory infections, including measles, vitamin A and its derivatives are reported to enhance the immune system and/or antibody response to virus vaccinations in children, particularly those with vitamin insufficiency. Retinoids are, therefore, proposed as an adjunct therapy in the treatment of COVID-19. The study is aimed to investigate the effects of vitamin A supplementation on disease improvement in pediatric and adolescent patients with either moderate or severe COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged between 1-month to 18-year old (boy or girl), 2) definitive or clinical diagnosis of severe acute respiratory syndrome (SARS)-like coronavirus 2 (SARS-COV-2) infection (by either a positive SARS-COV-2 polymerase chain reaction (PCR) test or a suggestive computed tomography (CT) scan, 3) no history or evidence of cancer or renal, hepatic, endocrine or viral disorders (including HIV/AIDS), 4) no history of supplementation either with vitamin A (VA) or with a multivitamin containing VA within the last 4 months, and 5) not participated in other clinical trials.

Exclusion Criteria:

* 1) mildly infected with SARS-COV-2 virus, and 2) pregnancy or lactation.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-21 (Estimated); Primary Completion 2021-11-21 (Estimated); Study Completion 2021-12-19 (Estimated)

PRIMARY OUTCOMES:
28-day mortality rate | within 28 days from end of intervention
  COVID-19 mortality rate is defined as the number of deaths per 100 pediatric COVID-19 cases 28 days from the date of the intervention.

SECONDARY OUTCOMES:
length of hospital stay | on the day of hospital discharge
  The length of hospital stay is defined as the difference between date of admission and date of discharge of the patient.
length of pediatric intensive care unit (PICU) stay | on the day of PICU discharge
  The length of PICU stay is defined as the difference between date of PICU admission and date of PICU discharge of the patient.
length of intubation | on the day of extubation
  The length of intubation is defined as the difference between date of beginning and end of intubation
length of mechanical ventilation | the weaning time of mechanical ventilation
  The length of mechanical ventilation is defined as the difference between date of beginning and end of mechanical ventilation.
multiple organ involvement | on the day of the particular organ involvement
  Multiple organ involvement is defined as one of either hematological, gastrointestinal, neurological, cardiovascular or hepatorenal complications.
complete blood count (CBC)/diff | before and within 3 days from end of intervention
  Complete blood count with differential
Prothrombin time (PT) | before and within 3 days from end of intervention
  Prothrombin time
Partial thromboplastin time (PTT) | before and within 3 days from end of intervention
  Partial thromboplastin time
International normalised ratio (INR) | before and within 3 days from end of intervention
  International normalised ratio
fibrinogen | before and within 3 days from end of intervention
  fibrinogen
troponin | before and within 3 days from end of intervention
  troponin
Aspartate transaminase (AST) | before and within 3 days from end of intervention
  Aspartate transaminase
Alanine transaminase (ALT) | before and within 3 days from end of intervention
  Alanine transaminase
Blood urea nitrogen (BUN) | before and within 3 days from end of intervention
  Blood urea nitrogen
Cr | before and within 3 days from end of intervention
  Creatinine
Erythrocyte sedimentation rate (ESR) | before and within 3 days from end of intervention
  Erythrocyte sedimentation rate
C-reactive protein (CRP) | before and within 3 days from end of intervention
  C-reactive protein
Lactate dehydrogenase (LDH) | before and within 3 days from end of intervention
  Lactate dehydrogenase
D-dimer | before and within 3 days from end of intervention
  D-dimer
ferritin | before and within 3 days from end of intervention
  ferritin
procalcitonin | before and within 3 days from end of intervention
  procalcitonin
vitamin A concentration | before and within 3 days from end of intervention
  vitamin A concentration

CONTACTS AND LOCATIONS:
Overall Officials: Seyede Sedigheh Hamzavi, MD, Principal Investigator — Professor Alborzi Clinical Microbiology Research Center, Shiraz University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No